CLINICAL TRIAL: NCT05034471
Title: Mi-STITCH™ and Mi-KNOT™ Device Technologies Improvement of Minimally Invasive Mitral Valve Repair - A Single-center, Pilot Clinical Safety & Feasibility Trial
Brief Title: Mi-STITCH™ and Mi-KNOT™ Device Technologies - Improvement of Mitral Valve Repair
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Collaborators: LSI SOLUTIONS, Inc. (Unknown)
Responsible Party: Principal Investigator, Martin Andreas, M.D., Assoc. Prof. PD Dr. Martin ANDREAS, MBA, PhD, MEBCTS, Medical University of Vienna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1228/2020
Record Dates: First submitted 2021-08-13; First posted 2021-09-05 (Actual); Last update posted 2021-12-08 (Actual); Status verified 2021-12

CONDITIONS: Mitral Regurgitation; Mitral Valve Insufficiency
Keywords: minimal invasive surgery; novel surgical device; mitral valve repair; cardiac surgery
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Mitral Valve Repair with Novel Device Technologies (Experimental): All study participants will undergo mitral valve repair by replacing the chordae tendinea with ePTFE single loop sutures using novel suturing devices.
  Interventions: Device: Mi-Chord™ Device Technologies

INTERVENTIONS:
Device: Mi-Chord™ Device Technologies — Mi-Chord™ System consists of LS-5™ ePTFE suture, the Mi-STITCH™ suturing device, the Mi-KNOT™ device and the Mi-KNOT™ titanium fastener. Mi-Chord™ system is designed to replace the chordae tendineae in order to enable mitral valve repair. These sub-devices (ePTFE suture, Mi-STITCH™, Mi-KNOT™ device, Mi-KNOT™ titanium fastener) can be considered as one system and refer to different aspects of the overall technology.

SUMMARY:
The objective of this study is to analyze the safety and efficacy of a novel device for minimally invasive mitral valve repair. Data of the early and intermediate postoperative period will be collected within routine clinical follow-up in order to assess morbidity and mortality as well as echocardiographic parameters.

DETAILED DESCRIPTION:
This study is a clinical, single-center pilot-study to evaluate safety and performance of a novel device in minimally invasive mitral valve surgery. Twelve (12) patients with mitral valve regurgitation planned for surgery at Vienna General Hospital (AKH) will be enrolled in the study considering inclusion and exclusion criteria. Mitral valve repair is achieved by replacing the chordae tendinea with expanded polytetrafluoroethylene (ePTFE) sutures either with or without concomitant procedures, such as annuloplasty, resection, or gap closure. These ePTFE sutures are placed between a mitral leaflet and the corresponding papillary muscle using a novel suturing device (Mi-Stitch™). By adjusting the length of the suture, the appropriate coaptation is achieved and prolapse is avoided - resulting in an adequate seal of the valve. The procedure will be assessed according to the primary safety endpoint (30 day mortality) as well as the implantation time. Likewise midterm safety endpoints at 12 months (mortality and observed rate of serious adverse events [SAE]) and procedural times will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Severe primary mitral valve regurgitation according to current guidelines with indication for mitral valve repair
* With or without concomitant procedures such as: coronary artery bypass grafting (CABG), other valve repair/replacement, pacemaker implantation, exclusion of left appendage and MAZE (or PVI) procedure, aortic procedures
* Euroscore II < 8
* Left ventricle ejection fraction > 35%
* Life expectancy above 1 year after the intervention based on operator assessment
* Willing to sign informed consent
* Willing to undergo all medical follow-ups necessary for the clinical investigations until study termination (echocardiography, blood tests, physical investigation)

Exclusion Criteria:

* Age <18 years
* Active endocarditis or myocarditis
* Previous cardiac surgery
* Heavily calcified mitral valve annulus
* Severe mitral stenosis
* Female pregnant patients
* Emergency procedures
* Patient not able to read or understand informed consent
* Patient not willing to sign informed consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2021-08-05 (Actual); Primary Completion 2022-03 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Primary safety endpoint - 30day Mortality | 30 days
  30 day Mortality
Primary efficacy endpoint - Implantation Time | intraoperative
  Defined as the period from start of valve assessment until the completion of the repair

SECONDARY OUTCOMES:
Secondary safety endpoints - Mortality | 1, 6 and 12 months
  Mortality
Secondary safety endpoints - Rate of SAEs | 1, 6 and 12 months
  Rate of serious adverse events according to the current EN ISO 14155 guidelines
Secondary efficacy endpoints - Procedural times | intraoperative
  Surgical time, aortic cross-clamp (ACC) time, cardiopulmonary bypass (CPB) time and time from first suture bite on mitral leaflet to final suture cutting and knot crimping on the papillary muscle (for each chord)

OTHER OUTCOMES:
Residual mitral valve regurgitation | 1 and 6 months
  Degree of mitral valve regurgitation (MR) at 1 and 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Andreas, MD, PhD, MBA, Principal Investigator — Department of Cardiac Surgery
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No